CLINICAL TRIAL: NCT05410366
Title: Safely Improving Emergency Diagnostic Testing Through Clinical Safe Harbors
Brief Title: Safe Harbors in Emergency Medicine, Specific Aim 3
Status: Withdrawn | Type: Observational
Why Stopped: Pursuing an alternative clinical trial
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alan Storrow, Associate Professor, Vanderbilt University Medical Center
Other Study IDs: AHRQ R18HS025931
Record Dates: First submitted 2022-06-02; First posted 2022-06-08 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-02

CONDITIONS: Low Back Pain; Headache; Head Injury, Minor
Keywords: Safe harbors; Emergency department; Liability
MeSH Terms: conditions — Low Back Pain; Headache; Craniocerebral Trauma; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Emergency department (ED) patients: Adult emergency department patients presenting with a chief complaint of 1) low back pain, 2) headache, or 3) minor head injury.
  Interventions: Other: Safe harbor clinical practice guideline

INTERVENTIONS:
Other: Safe harbor clinical practice guideline — A safe harbor is a special type of clinical practice guideline which, under existing federal law, may serve as the legal standard of care, not just evidence of the standard of care. If a patient with a safe harbor condition satisfies all safe harbor inclusion criteria and does not meet any exclusion criteria, no imaging is required, and the patient may be discharged with specific instructions. If a patient is excluded from the safe harbor, then imaging decisions are per customary practice. The safe harbor clinical practice guidelines are provided to treating ED physicians, but they are not obligated to use them. The safe harbor pathways do not limit the diagnostic and therapeutic approach patients and physicians undertake during a clinical encounter. They have the liberty in this decision to proceed jointly down a clinical pathway most appropriate to the individual clinical circumstance.

SUMMARY:
Many patients who present to the emergency department (ED) receive a vast array of diagnostic tests, some of which might not be useful. Providers often feel obligated to order so many tests to protect themselves against the risk of being sued. The investigators believe if a standard of care providing legal protection for certain clinical conditions were agreed upon and followed, unnecessary testing would significantly decrease in the ED, which, in turn, would improve patient safety, augment the quality of care delivered, and increase patient satisfaction.

DETAILED DESCRIPTION:
Overutilization of healthcare resources often has negative implications. The Choosing Wisely campaign, an initiative of the American Board of Internal Medicine, was proposed to help patients and caregivers engage in shared conversations to reduce overuse of potentially harmful tests and procedures. However, the Choosing Wisely campaign's lack of linkage to medical liability considerations has substantially reduced its impact.

For instance, excessive medical imaging and its associated radiation exposure inflicts a measurably real and significant risk of carcinogenesis, drives costs, and therefore is a significant Choosing Wisely target. This is a particularly important consideration in the emergency care setting, frequently cited as an extremely utilization rich environment due to the higher inherent risk of missed pathology and the isolation of clinical care.

The investigators hypothesize a special type of predetermined standard of care (a "safe harbor") can be defined based upon medical evidence, and upon consultation among multiple experts and advisors, for a selected number of clinical conditions within the specialty of emergency medicine (EM). Furthermore, a state-based, federally-contracted and legally-recognized Quality Improvement Organization (QIO) could adopt the "safe harbor" and, in doing so, establish the standard of care in the context of a legal liability claim. Practitioners who meet such a standard and implement it appropriately satisfy their obligation under the law of medical malpractice.

Ultimately, defining provider liability through this predetermined, or ex ante, standard of care, may result in a significant reduction in healthcare resource utilization within EM. Through this reduction, the quality of care would not decrease and a measurable reduction in radiation exposure would occur. Moreover, these predefined standards of care would improve communication between patient and provider during the clinical transaction.

A team of Vanderbilt University medicine, law, economics, and clinical faculty will undertake this. The investigators have summoned a broad group of technical experts and advisors and defined safe harbors for a narrow set of distinct clinical conditions within EM. These safe harbors will be presented for review and approval by the appropriate QIO. Specific Aim 3 will advance the safe harbor demonstration to EM practitioners at Vanderbilt University Medical Center and determine the effects on radiation exposure, length of stay, patient satisfaction, patient costs, charges, and adverse event reporting.

ELIGIBILITY:
Inclusion Criteria:

* Adult emergency department patients presenting with a chief complaint of 1) low back pain, 2) headache, or 3) minor head injury.

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Vanderbilt University Medical Center emergency department patients. Comparator Northwestern University emergency department patients.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Radiation exposure | June 15, 2022 - March 31, 2024
  Aggregate ED radiologic imaging - X-ray or CT scan and MRI

SECONDARY OUTCOMES:
Length of stay | June 15, 2022 - March 31, 2024
  Aggregate ED length of stay defined as provider evaluation to disposition

OTHER OUTCOMES:
Patient satisfaction | June 15, 2022 - March 31, 2024
  Press Ganey scores, Consumer Assessment of Healthcare Providers and Systems (CAHPS), aggregate number of patient complaints
Patient cost | June 15, 2022 - March 31, 2024
  Aggregate out of pocket patient costs
Patient charges | June 15, 2022 - March 31, 2024
  Aggregate patient charges
Adverse event reporting | June 15, 2022 - March 31, 2024
  Aggregate number of reports per patient per condition

CONTACTS AND LOCATIONS:
Overall Officials: Alan B Storrow, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blumstein JF, McMichael BJ, Storrow AB. Constraints on Medical Liability Through Malpractice Safe Harbors. JAMA Health Forum. 2020;1(8):e200961. doi: 10.1001/jamahealthforum.2020.0961. Epub 2020 Aug 14. No abstract available. PMID 33728420